CLINICAL TRIAL: NCT00450957
Title: Phase I Multiple Dose Pharmacokinetic Study of the Dietary Supplement Lycopene Delivered in Capsule Form to Healthy Male Volunteers Between 18 and 55 Years of Age
Brief Title: Lycopene in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2012-02709; UIC-2006-0853; CDR0000536181; N01CN85081 (Other Grant/Funding Number: US NIH Grant/Contract Award Number)
Record Dates: First submitted 2007-03-20; First posted 2007-03-22 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2013-04

CONDITIONS: Healthy, no Evidence of Disease; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Lycopene

ARMS (2):
- Arm I (high-dose lycopene) (Experimental): Participants receive high-dose oral lycopene once or twice a day for 14 days. After 2 weeks of a lycopene-free period, participants crossover and receive high-dose lycopene at the alternative daily schedule (once or twice a day) for 14 days.
  Interventions: Dietary Supplement: lycopene; Other: pharmacological study
- Arm II (low-dose lycopene) (Experimental): Participants receive low-dose oral lycopene once or twice a day for 14 days. After 2 weeks of a lycopene-free period, participants crossover and receive low-dose lycopene at the alternative daily schedule (once or twice a day) for 14 days
  Interventions: Dietary Supplement: lycopene; Other: pharmacological study

INTERVENTIONS:
Dietary Supplement: lycopene — Given orally
  Other Names: all-trans-Lycopene; Lyc-O-Mato; LYCO; psi,psi-Carotene
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This randomized phase I trial is studying the side effects and best dose of lycopene in healthy male participants. Chemoprevention is the use of certain drugs to keep cancer from forming. The use of lycopene, a substance found in tomatoes, may prevent prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Compare the toxicity and safety of 2 different doses of oral lycopene in healthy male participants.

II. Compare the pharmacokinetics of 2 different doses of this drug in these participants.

III. Determine the toxicity and pharmacokinetics needed to proceed to a large phase II/III study in men at high risk for prostate cancer.

OUTLINE: This is a randomized, crossover study. Participants are randomized to 1 of 2 treatment arms.

Arm I: Participants receive high-dose oral lycopene once or twice a day for 14 days. After 2 weeks of a lycopene-free period, participants crossover and receive high-dose lycopene at the alternative daily schedule (once or twice a day) for 14 days.

Arm II: Participants receive low-dose oral lycopene once or twice a day for 14 days. After 2 weeks of a lycopene-free period, participants crossover and receive low-dose lycopene at the alternative daily schedule (once or twice a day) for 14 days.

Treatment continues in the absence of unacceptable toxicity. Participants adhere to dietary restrictions for 2 weeks at baseline, 2 weeks during study treatment, and 2 weeks during pharmacokinetic sampling.

Blood samples are collected periodically at baseline and during study treatment for pharmacokinetic studies.

PROJECTED ACCRUAL: A total of 20 participants will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers judged to be in good medical condition based on history and physical exam
* Karnofsky performance status 100%
* AST and ALT ≤ 75 IU/L
* Bilirubin ≤ 2.0 mg/dL
* Creatinine ≤ 1.5 mg/dL
* Hemoglobin ≥ 13.0 g/dL
* WBC ≥ 4,000/mm³
* Platelet count ≥ 150,000/mm³ and ≤ 400,000/mm³
* Must be within height and weight standards identified by Metropolitan Life scales
* Nonsmoker (for ≥ 3 months)
* No history of alcohol abuse
* No history of gastrointestinal malabsorption or other condition that could affect drug absorption
* No history of a psychiatric condition
* No chronic medical condition
* No active history of any of the following:

  * Cancer
  * Liver disease
  * Cardiovascular disease
  * Renal disease
  * Diabetes mellitus
  * Other illnesses that, in the opinion of the investigator, could represent a threat for the participants life
* No allergy to tomato-based products
* No lycopene in the diet for ≥ 14 days
* At least 4 weeks since prior and no other concurrent experimental medications
* No concurrent participation in another experimental study
* No concurrent use of regular prescription medication or over-the-counter medications
* No concurrent vitamin, mineral, or herbal supplements

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2006-10; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Toxicity according to NCI Common Toxicity Criteria (CTC) version 3.0 | 2 weeks
Safety according to NCI CTC version 3.0 | 12 weeks
Pharmacokinetics | At baseline, at 12, 24, 36, 48, 72, 96, 120, 168, 216, 288, and 360 hours

CONTACTS AND LOCATIONS:
Overall Officials: Keith Rodvold, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois, Chicago, Illinois, United States